CLINICAL TRIAL: NCT03955120
Title: Validation of the Dayzz Digital Sleep Training App in Insomnia and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dayzz Live Well Ltd. (Industry)
Collaborators: Israel Innovation Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dayzz_002
Record Dates: First submitted 2019-02-07; First posted 2019-05-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Insomnia; Sleep Apnea
Keywords: sleep disorders; cognitive and behavioral treatment; digital treatment; insomnia; sleep apnea; sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes; Sleep Wake Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Apnea- Dayzz (Experimental): The intervention group is also provided access to the dayzz app, a personalized digital sleep training program. The sleep training begins a sleep assessment questionnaire and ongoing sleep and activity data collection which is used to tailor an individualized sleep training program including behavioral and cognitive techniques to improve the adherence to CPAP. The dayzz sleep program is composed of three main components, (1) a mobile digital program via the dayzz app, (2) guidance of a sleep trainer, and (3) an ambulatory sleep monitoring device. The intervention group meets a CPAP technician at the sleep clinic, as detailed below in the Sleep Apnea TAU group
  Interventions: Behavioral: Dayzz mobile sleep training
- Sleep Apnea- Treatment as Usual (Active Comparator): The "treatment as usual" [TAU] group meets a CPAP technician at the sleep clinic, who provides the participant with a CPAP device and fits the mask. The will also receive a follow-up visit with the same technician for technical support, mask changes or alterations if needed after an initial 7 to 14-day at home CPAP trial.
  Interventions: Other: Treatment as usual
- Insomnia - Dayzz (Experimental): The intervention group is provided access to the dayzz app, a personalized digital sleep training program. The sleep training begins a sleep assessment questionnaire and ongoing sleep and activity data collection which is used to tailor an individualized sleep training program including behavioral and cognitive techniques to improve the insomnia concerns, sleep symptoms, and achieve sleep goals. The dayzz sleep program is composed of three main components, (1) a mobile digital program via the dayzz app, (2) guidance of a sleep trainer, and (3) an ambulatory sleep monitoring device.
  Interventions: Behavioral: Dayzz mobile sleep training
- Insomnia - Treatment as Usual (Active Comparator): The "treatment as usual" [TAU] group, will receive standard treatment recommendations for their insomnia, including sleep hygiene suggestions, referral for supportive/non-medical treatments [e.g. relaxation therapies], and if needed hypnotics or other medications prescribed by the sleep clinic physician.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Dayzz mobile sleep training — 1. The dayzz digital sleep program provides each user with relevant educational materials (depending on their sleep condition), sleep tracking, and sleep or health-related tasks or challenges pertaining to their sleep or sleep difficulties.
  2. Each app user is matched with a "sleep trainer" who will communicate with them via a "chat" option within the dayzz app and who will support the participants with any sleep training issues or technical aspects of all app for the duration of the treatment program.
  3. Participants receive a wrist-worn device for monitoring sleep and activity patterns, a Fitbit fitness tracker (www.fitbit.com), to be worn for the duration of the study.
  Arms: Insomnia - Dayzz; Sleep Apnea- Dayzz
Other: Treatment as usual — Standard medical care for specific sleep condition
  Arms: Insomnia - Treatment as Usual; Sleep Apnea- Treatment as Usual

SUMMARY:
The prevalence of sleep disorders has achieved epidemic proportions in Western countries. Despite this, assessment and treatment of sleep disorders remains infrequent, unattainable, and often costly. Dayzz is aware of the need for easily accessible, user-friendly, and affordable treatment strategies for known sleep conditions. This research proposes a randomized controlled outcome study aimed to validate a, digitized, cost-effective mobile app which assesses and manages insomnia and CPAP adherence in persons with sleep apnea. The app's sleep training protocols recommend life-style and behavioral changes and tracks these changes with the aim of improving sleep and well-being. In this study, the dayzz app digital treatment protocol will be compared to the standard treatment for these sleep conditions by a sleep professional.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-65 years of age referred to the Carmel Hospital sleep clinic and diagnosed by the clinic physician with either Sleep Apnea (referred for CPAP treatment) or Insomnia.

Exclusion Criteria:

* Patient age <21 years.
* Patient who is not a member of Clalit Healthcare services.
* Persons with insufficient control of the English language required for adequate use of app.
* Persons with insufficient experience/knowledge and/or use of digital apps/smartphones.
* Persons with serious medical or psychiatric conditions.
* Women who are pregnant or breastfeeding.
* Nighttime shift-workers.
* Persons who are unable to provide consent due to mental incapacity.
* Persons referred for evaluation of sleep by Ministry of Transportation (for licensing purposes).
* Persons with comorbid insomnia and sleep apnea

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Total sleep time (minutes) | 3 months to 1 year
  sleep duration in minutes per night (based on nightly sleep diary)
Sleep onset latency (minutes) | 3 months to 1 year
  Number of minutes to fall asleep per night (based on nightly sleep diary)
Wake after sleep onset (minutes) | 3 months to 1 year
  Number of minutes awake in total per night (based on nightly sleep diary)
Sleep efficiency (percent) | 3 months to 1 year
  (Number of minutes asleep per night/number of minutes in bed per night)*100 (based on sleep diary data)
Sleep quality | 3 months to 1 year
  Likert scale of sleep quality between 1 and 10 (based on sleep diary report)
Nightly CPAP use | 3 months to 1 year
  Minutes of wearing the CPAP mask per night (based on sleep diary report)
Excessive daytime sleepiness | 3 months to 1 year
  The Epworth Sleepiness Scale (ESS): The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity or their 'daytime sleepiness'.
Sleep symptom screening questionnaire | 3 months to 1 year
  The Dayzz Sleep Questionnaire is a digitized screening measure that assesses sleep quantity and quality and presence/risk for specific sleep disorders. It is composed of some self-rated items, assessing sleep amounts, sleep quality, excessive sleepiness, and risk factors for sleep-related breathing disorders, symptoms of insomnia and sleep/wake circadian rhythms. The questions are based on the International Classification of Sleep Disorders (3rd Edition; American Academy of Sleep Medicine) diagnostic criteria for four common categories of sleep disorders: Insomnia, Insufficient Sleep Syndrome, Sleep Apnea Disorders, and Circadian Rhythm Sleep-Wake Disorders.
Insomnia severity | 3 months to 1 year
  The Insomnia Severity Index (ISI) is a well-validated 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia over the past month (Morin, 1993). The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

SECONDARY OUTCOMES:
Work productivity | 3 months to 1 year
  The Work Productivity and Activity Impairment Questionnaire-Specific Health problem (WPAI:SHP): The WPAI is a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to a specific health problem (Reilly et al, 1993). WPAI:SHP outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Insomnia-related quality of life | 3 months to 1 year
  The Glasgow Sleep Impact Index (GSII). Administered only to the insomnia sample. The GSII is a self-report measure which asks patients to generate, and assess, three domains of measure insomnia-related quality of life impairment. These three patient-generated areas of impairment are ranked in order of concern (1-3; i.e. 1=the most concerning impairment), and then rated on a visual analogue scale with respect to impact in the past two weeks. Patients re-rate these specified areas of impairment, post-intervention, permitting both individual and group-level analyses.
Sleep Apnea-related Quality of Life-Short form (SAQLI-SF) | 3 months to 1 year
  The SAQLI- SF (for sleep apnea sample only) measures the effects of sleep apnea on a person's quality of life. The questions represent four quality of life domains: Daily Activities, Social Interactions, Emotions,and Symptoms. Two total scores will be generated, which reflect the pre- and post-treatment quality of life. The total scores range between 1-14, with higher values representing poorer outcomes. No subscale scores are generated.
The WHO-5 Well-being Index (WHO-5) | 3 months to 1 year
  The WHO-5 Well-being Index (WHO-5) is a short, self-administered questionnaire measuring psychological well-being. It covers 5 positively worded items, related to positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interests (being interested in things). Each of the five items is rated on a 6-point Likert scale from 0 (= not present) to 5 (= constantly present). Scores are summated, with raw score ranging from 0 to 25. Then the scores are transformed to 0-100 by multiplying by 4 which provides the total score, with higher scores meaning better well-being. The scale does not generate subscale scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Hospital, Haifa, Israel